CLINICAL TRIAL: NCT03700229
Title: An Open-label Phase II Study to Determine the Efficacy and Safety of Rituximab and Bortezomib in Patients With Newly Diagnosed Acquired Hemophilia A
Brief Title: Study to Evaluate Rituximab and Bortezomib in Patients With Newly Diagnosed Acquired Hemophilia A
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Tienan Zhu, Associate chief physician, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-AHA-001
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Acquired Hemophilia A
MeSH Terms: conditions — Factor 8 deficiency, acquired | interventions — Bortezomib; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bortezomib +Rituximab (Experimental): Bortezomib +Rituximab
  Interventions: Drug: Bortezomib; Drug: Rituximab

INTERVENTIONS:
Drug: Bortezomib — Bortezomib intravenously 1.3mg/m2 d1,4,8,11 for 4 doses
Drug: Rituximab — rituximab intravenously 500 mg for one dose

SUMMARY:
The purpose of this prospective study is to determine the efficacy and safety of Rituximab plus Bortezomib in patients with newly diagnosed acquired hemophilia A.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label clinical trial to evaluate the efficacy and safety the regimen of Bortezomib with rituximab as first-line treatment to eradicate anti-factor VIII antibodies in newly diagnosed acquired hemophilia A.

All of enrolled patients in this study will be injected Bortezomib plus rituximab. This study will be performed for about 2 years and approximately 22 patients will be enrolled in our insititution.

After obtaining the written informed consent from the patients, the information of demographic and medical history will be collected and laboratory tests will be performed.

Patients who meet the inclusion/exclusion criteria will be received the regimens: Bortezomib (1.3mg/m2 d1,4,8,11) with rituximab (375mg/m2 for one dose). The information of adverse events will be collected. In case that the evaluation of treatment response might be performed in regular clinical practice, those data will also be collected as well.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥ 18 years;
2. Understand and voluntarily sign an ICD prior to any study related assessments/procedures are conducted;
3. Diagnosis of acquired hemophilia A；
4. acute bleeding episodes(≥once).

Exclusion Criteria:

1. Uncontrolled systemic infection;
2. Allergy to rituximab;
3. Positive for Lupus anticoagulant;
4. Life expectancy < 3 months;
5. Pregnant and breastfeeding women;
6. Neuropathy>Grade 1;
7. Positive for Hepatitis B surface antigen or hepatitis C antibody or human immunodeficiency virus（HIV）antibody;
8. Patients with poor compliance；
9. Patient who is considered by the investigator not suitable for clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2020-04-15 (Estimated)

PRIMARY OUTCOMES:
The time to attain first complete remission (CR) | Last day of the treatment regimen (up to 3 months)
  Complete remission defined as titer FVIII inhibitor lower than 0.6 Bethesda unit, factor VIII level> 50% and no bleeding events without bypass treatments for 24 hours

SECONDARY OUTCOMES:
The time to durable treatment response | During 24 month
  The time to durable treatment response was defined as the time from date of achieving CR until the date of relapse or date of death from any cause（whichever came first）
Adverse events | During 24 month
  Include major bleeding, infection, nerve toxicity, and so on.
Overall survival | During 24 month
  Overall survival was defined as the time from date of first diagnosis until the date of death from any cause，and death from any cause will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tienan Zhu, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Collins P, Baudo F, Knoebl P, Levesque H, Nemes L, Pellegrini F, Marco P, Tengborn L, Huth-Kuhne A; EACH2 registry collaborators. Immunosuppression for acquired hemophilia A: results from the European Acquired Haemophilia Registry (EACH2). Blood. 2012 Jul 5;120(1):47-55. doi: 10.1182/blood-2012-02-409185. Epub 2012 Apr 18. PMID 22517903
- [Background] Bras GP, Pinto RJ, Carvalho MM, Fernandes SP, Andrade JJ, Guimaraes JE. Bortezomib: Potential Key Role in the Treatment of Multiple Myeloma-Related Acquired Hemophilia A. Semin Thromb Hemost. 2017 Feb;43(1):109-112. doi: 10.1055/s-0036-1597648. Epub 2016 Dec 19. No abstract available. PMID 27992938
- [Background] Bonfanti C, Crestani S, Frattini F, Sissa C, Franchini M. Role of rituximab in the treatment of postpartum acquired haemophilia A: a systematic review of the literature. Blood Transfus. 2015 Jul;13(3):396-400. doi: 10.2450/2014.0242-14. Epub 2014 Dec 17. No abstract available. PMID 25545867
- [Result] Ratnasingam S, Walker PA, Tran H, Kaplan ZS, McFadyen JD, Tran H, Teh TC, Fleming S, Catalano JV, Chunilal SD, Johnston A, Opat SS, Shortt J. Bortezomib-based antibody depletion for refractory autoimmune hematological diseases. Blood Adv. 2016 Nov 22;1(1):31-35. doi: 10.1182/bloodadvances.2016001412. eCollection 2016 Nov 29. PMID 29296693